CLINICAL TRIAL: NCT05177666
Title: Patients With Advanced Refractory Solid Tumors Who Failed Standard Treatments and Matched Individualized Treatment Based on Tumor Molecular Characteristics: a Prospective Registration Study
Brief Title: a Prospective Registration Study for Patients With Advanced Refractory Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Collaborators: Tianjin Happy Life Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: V1
Record Dates: First submitted 2021-11-24; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Feasibility; Effectiveness; Safety; Targeted Molecular Therapy
MeSH Terms: interventions — Trastuzumab; pertuzumab; Vemurafenib; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The patient undergoes biopsy sampling for next-generation sequencing (NGS) testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Targeted therapy — Based on next-generation sequencing (NGS) detection, after discussion by the Molecular Steering Committee (MTB), intervention guidance suggestions are given based on domestic and foreign guidelines and clinical experience, and finally the patient and clinician jointly choose the treatment plan.
  Other Names: Entratinib; Cabotinib; Aletinib; Enmetrastuzumab; Trastuzumab; Pertuzumab; Vemurafenib; Atilizumab; Bevacizumab; Erlotizumab

SUMMARY:
This is a prospective registration study for patients with advanced refractory solid tumors. Patients who meet the eligibility criteria will be included to participate in the study, and baseline information to be collected after signed informed consent. Patients will choose for themselves whether to carry out targeted therapy or other appropriate treatment methods. And we plan to follow up for at least 12 months or until disease progression or death.

DETAILED DESCRIPTION:
1. Screen and enroll 120 patients with refractory solid tumors, and sign informed consents;
2. Extract the clinical data, including gender, age, disease diagnosis, past treatment history and genetic test results, etc.;
3. Take biopsy samples and perform NGS testing on patients. After discussion by the Molecular Steering Committee (MTB), the recommendations for treatment guidance will be given based on treatment guidelines and clinical experience;
4. The patient and the clinician jointly select the treatment plan and follow-up until the patient's disease progresses. The follow-up time will be 1 year;
5. During the follow-up period, clinical treatment and routine examination information of patients will be collected;
6. If the patient fails to receive molecular targeted therapy or they cannot tolerate the adverse reaction of the drug after adequate treatment, the clinician will evaluate whether a second NGS resistance test is needed or the participant may withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic malignant solid tumor confirmed by histology or cytology
* Disease progression or intolerance after receiving standard treatment
* With evaluable lesions (RECIST 1.1 standard)
* Tumor tissue pieces with sufficient formalin-fixed paraffin-embedded (FFPE) can be used for genetic testing
* ECOG PS score 0-4 (3-4 points only for patients with tumor burden)
* Sign the informed consent form

Exclusion Criteria:

* The subject is participating in any other clinical research;
* Researchers believe that serious or uncontrolled medical diseases (ie uncontrolled diabetes, chronic kidney disease, chronic lung disease, or uncontrolled active infections, mental illnesses/social conditions that restrict compliance with research requirements) that will confuse the analysis of research treatment response ；
* Patients during pregnancy or lactation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From November 2021 to November 2022, the patients with refractory tumors who underwet the standard treatment standard treatment, went to the Shenzhen Hospital of the University of Hong Kong and were willing to have genetic testing for individualized targeted therapy. It is planned to enroll 120 patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2021.11-2023.11
  ORR is judged based on RECIST 1.1 criteria for all treatment groups at each visit period.
Proportion of targeted therapy guided by tumor molecular characteristics | 2021.11-2023.11
  The proportion of all enrolled patients receiving targeted therapy guided by tumor molecular characteristics during the study period, would be calculated, which defined as having received one or more the treatments based on tumor molecular characteristics.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2021.11-2023.11
  PFS is defined as the time from the first administration to disease progression or death.
Overall survival (OS) | 2021.11-2023.11
  OS is defined as the time from the first administration to death from any cause.
Best overall response (BOR) | 2021.11-2023.11
  The effectiveness of a patient would be evaluated multiple times, and the best one is defined as the best overall response.
Adverse events | 2021.11-2023.11
  The incidence of serious adverse events in each group, which is judged based on CTCAE v5.0 standard.
Quality of Life Score (QoL) | 2021.11-2023.11
  The QoL is evaluated by the scale (0PROMIS-29 Profile v2.1) at each visit period for all the enrolled patients.
Proportion of patients with intervening genomic variants | 2021.11-2023.11
  The intervening genomic variants are defined by the conclusion after MTB discussion.

OTHER OUTCOMES:
Changes in ECOG score before and after treatment | 2021.11-2023.11
  We compare the ECOG scores of each visit with the baseline, including the number and proportion, and the difference.
Proportion of targeted therapy guided by second tumor molecular characteristics | 2021.11-2023.11
  After targeted therapy drug resistance, then the proportion of targeted therapy guided by the second tumor molecular characteristics would be calculated during study period.

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Li, MD, Principal Investigator — The University of Hong Kong-Shenzhen Hospital; Weitang Wu, Principal Investigator — The University of Hong Kong-Shenzhen Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gerlinger M, Rowan AJ, Horswell S, Math M, Larkin J, Endesfelder D, Gronroos E, Martinez P, Matthews N, Stewart A, Tarpey P, Varela I, Phillimore B, Begum S, McDonald NQ, Butler A, Jones D, Raine K, Latimer C, Santos CR, Nohadani M, Eklund AC, Spencer-Dene B, Clark G, Pickering L, Stamp G, Gore M, Szallasi Z, Downward J, Futreal PA, Swanton C. Intratumor heterogeneity and branched evolution revealed by multiregion sequencing. N Engl J Med. 2012 Mar 8;366(10):883-892. doi: 10.1056/NEJMoa1113205. PMID 22397650
- [Result] Hoadley KA, Yau C, Wolf DM, Cherniack AD, Tamborero D, Ng S, Leiserson MDM, Niu B, McLellan MD, Uzunangelov V, Zhang J, Kandoth C, Akbani R, Shen H, Omberg L, Chu A, Margolin AA, Van't Veer LJ, Lopez-Bigas N, Laird PW, Raphael BJ, Ding L, Robertson AG, Byers LA, Mills GB, Weinstein JN, Van Waes C, Chen Z, Collisson EA; Cancer Genome Atlas Research Network; Benz CC, Perou CM, Stuart JM. Multiplatform analysis of 12 cancer types reveals molecular classification within and across tissues of origin. Cell. 2014 Aug 14;158(4):929-944. doi: 10.1016/j.cell.2014.06.049. Epub 2014 Aug 7. PMID 25109877
- [Result] Ciriello G, Miller ML, Aksoy BA, Senbabaoglu Y, Schultz N, Sander C. Emerging landscape of oncogenic signatures across human cancers. Nat Genet. 2013 Oct;45(10):1127-33. doi: 10.1038/ng.2762. PMID 24071851
- [Result] Wheler J, Lee JJ, Kurzrock R. Unique molecular landscapes in cancer: implications for individualized, curated drug combinations. Cancer Res. 2014 Dec 15;74(24):7181-4. doi: 10.1158/0008-5472.CAN-14-2329. Epub 2014 Oct 17. PMID 25326492
- [Result] Von Hoff DD, Stephenson JJ Jr, Rosen P, Loesch DM, Borad MJ, Anthony S, Jameson G, Brown S, Cantafio N, Richards DA, Fitch TR, Wasserman E, Fernandez C, Green S, Sutherland W, Bittner M, Alarcon A, Mallery D, Penny R. Pilot study using molecular profiling of patients' tumors to find potential targets and select treatments for their refractory cancers. J Clin Oncol. 2010 Nov 20;28(33):4877-83. doi: 10.1200/JCO.2009.26.5983. Epub 2010 Oct 4. PMID 20921468
- [Result] Tsimberidou AM, Iskander NG, Hong DS, Wheler JJ, Falchook GS, Fu S, Piha-Paul S, Naing A, Janku F, Luthra R, Ye Y, Wen S, Berry D, Kurzrock R. Personalized medicine in a phase I clinical trials program: the MD Anderson Cancer Center initiative. Clin Cancer Res. 2012 Nov 15;18(22):6373-83. doi: 10.1158/1078-0432.CCR-12-1627. Epub 2012 Sep 10. PMID 22966018
- [Result] Schwaederle M, Parker BA, Schwab RB, Daniels GA, Piccioni DE, Kesari S, Helsten TL, Bazhenova LA, Romero J, Fanta PT, Lippman SM, Kurzrock R. Precision Oncology: The UC San Diego Moores Cancer Center PREDICT Experience. Mol Cancer Ther. 2016 Apr;15(4):743-52. doi: 10.1158/1535-7163.MCT-15-0795. Epub 2016 Feb 12. PMID 26873727
- [Result] Le Tourneau C, Delord JP, Goncalves A, Gavoille C, Dubot C, Isambert N, Campone M, Tredan O, Massiani MA, Mauborgne C, Armanet S, Servant N, Bieche I, Bernard V, Gentien D, Jezequel P, Attignon V, Boyault S, Vincent-Salomon A, Servois V, Sablin MP, Kamal M, Paoletti X; SHIVA investigators. Molecularly targeted therapy based on tumour molecular profiling versus conventional therapy for advanced cancer (SHIVA): a multicentre, open-label, proof-of-concept, randomised, controlled phase 2 trial. Lancet Oncol. 2015 Oct;16(13):1324-34. doi: 10.1016/S1470-2045(15)00188-6. Epub 2015 Sep 3. PMID 26342236
- [Result] Abrahams E, Eck SL. Molecular medicine: Precision oncology is not an illusion. Nature. 2016 Nov 17;539(7629):357. doi: 10.1038/539357e. No abstract available. PMID 27853199
- [Result] Mosele F, Remon J, Mateo J, Westphalen CB, Barlesi F, Lolkema MP, Normanno N, Scarpa A, Robson M, Meric-Bernstam F, Wagle N, Stenzinger A, Bonastre J, Bayle A, Michiels S, Bieche I, Rouleau E, Jezdic S, Douillard JY, Reis-Filho JS, Dienstmann R, Andre F. Recommendations for the use of next-generation sequencing (NGS) for patients with metastatic cancers: a report from the ESMO Precision Medicine Working Group. Ann Oncol. 2020 Nov;31(11):1491-1505. doi: 10.1016/j.annonc.2020.07.014. Epub 2020 Aug 24. PMID 32853681